CLINICAL TRIAL: NCT02479490
Title: Phase II Study of Oral PRednisone 5 mg Bid Plus EVerolimus in Patients With Metastatic Renal Cell Cancer After Failure of Vascular Endothelial Growth Factor Receptor-tyrosine Kinase Inhibitors
Brief Title: PRednisone Plus EVerolimus in Patients With Metastatic Renal Cell Cancer After Failure of VEGFR -TKI
Acronym: PREV
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Istituto Romagnolo per lo Studio dei Tumori Dino Amadori IRST S.r.l. IRCCS (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRST189.04
Record Dates: First submitted 2015-06-19; First posted 2015-06-24 (Estimated); Last update posted 2018-01-16 (Actual); Status verified 2018-01

CONDITIONS: Metastatic Renal Cancer
Keywords: metastatic renal cancer; failure of VEGFR_TKI; prednisone; everolimus
MeSH Terms: conditions — Kidney Neoplasms | interventions — Prednisone; Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Prednisone + Everolimus (Experimental): Prednisone + Everolimus
  Interventions: Drug: Prednisone + Everolimus

INTERVENTIONS:
Drug: Prednisone + Everolimus — Prednisone + Everolimus: Everolimus is formulated as tablets of 5-10 mg strength, blister-packed under aluminium foil in units of 10 tablets. Prednisone will be dispensed to patients at the dose of 5 mg twice daily (BID). Everolimus at dose of 10 mg (one 10 mg tablet or two 5 mg tablets). Both drugs will be self-administered orally, continuously from Day 1 (Visit 2) until progression of disease, unacceptable toxicity, death or discontinuation for any other reason.
  A treatment cycle consists of 28 days.
  Other Names: prednisone; everolimus

SUMMARY:
This is a multicenter prospective study that includes all patients with metastatic Renal Cell Cancer (RCC) pre- treated with VEGFR TKI in eight Italian cancer centers.

Everolimus is formulated as tablets of 5-10 mg strength, blister-packed under aluminium foil in units of 10 tablets. Prednisone will be dispensed to patients at the dose of 5 mg twice daily (BID). Everolimus at dose of 10 mg (one 10 mg tablet or two 5 mg tablets). Both drugs will be self-administered orally, continuously from Day 1 (Visit 2) until progression of disease, unacceptable toxicity, death or discontinuation for any other reason.

A treatment cycle consists of 28 days.

DETAILED DESCRIPTION:
Title Phase II study of oral PRednisone 5 mg bid plus EVerolimus in patients with metastatic renal cell cancer after failure of vascular endothelial growth factor receptor-tyrosine kinase inhibitor (PREV study).

Short Title/ Acronym PREV Protocol Code IRST189.04 Phase Phase 2 Study Design This is a multicenter prospective study that includes all patients with metastatic RCC pre- treated with VEGFR TKI in eight Italian cancer centers.

Study Duration 2 years of recruitment and 1 year of follow-up Study Center(s) multi-center: 8 centers involved

Objectives Primary objective:

To evaluate the safety and tolerability of prednisone 5 mg bid and everolimus 10 mg/day in RCC.

Secondary objectives:

To evaluate the activity and the clinical outcome of these patients.

Exploratory objectives:

To evaluate the influence of prednisone on trough concentration of everolimus and correlation with the incidence of side effects, in particular stomatitis and non-infectious pneumonitis.

Infiammation markers such as pentraxin 3 (PTX3), IL-6, TGF-β and neutrophil-lymphocyte ratio will be correlated with clinical outcome (ORR, PFS, OS).

Number of Subjects 42 subjects Diagnosis and Main Inclusion Criteria Patients with mRCC who failed at least one VEGFR TKI.

Main Inclusion Criteria:

* Patients with renal cell carcinoma who failed at least one VEGFR TKI
* Patients with adequate bone marrow function
* Patients with adequate liver function
* Patients with adequate renal function Diagnosis and Main Inclusion Criteria (continued) Main exclusion criteria:
* CNS disease OR patients with presence or history of central nervous system (CNS) lymphoma
* Patients receiving chronic, systemic treatment with corticosteroids or another immunosuppressive agent (except corticosteroids with a daily dosage equivalent to prednisone ≤ 20 mg for adrenal insufficiency). However, patients receiving corticosteroids must be on a stable dose for ≥ 4 weeks prior to the first dose of everolimus. Topical or inhaled corticosteroids are permitted.
* Patients with a known hypersensitivity to everolimus or other rapamycins (sirolimus, temsirolimus) or to its excipients
* Patients with uncontrolled hyperlipidemia (≥ Grade 3 hyperlipidemia despite optimal supportive medical therapy)
* Patients with an active, bleeding diathesis
* Previous organ transplantation
* Patients who have any severe and/or uncontrolled medical conditions or other conditions that could affect their participation in the study Study Product, Dose, Route, Regimen and duration of administration Everolimus is formulated as tablets of 5-10 mg strength, blister-packed under aluminium foil in units of 10 tablets. Prednisone will be dispensed to patients at the dose of 5 mg twice daily (BID). Everolimus at dose of 10 mg (one 10 mg tablet or two 5 mg tablets). Both drugs will be self-administered orally, continuously from Day 1 (Visit 2) until progression of disease, unacceptable toxicity, death or discontinuation for any other reason.

A treatment cycle consists of 28 days. Reference therapy Not applicable Statistical Methodology This is a multicenter prospective study that includes all patients with metastatic RCC pre- treated with VEGFR TKI in eight Italian cancer centers.

The study will be analyzed on an intent-to-treat basis. Secondary parameters will be analyzed exploratively for the intent-to-treat population.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old
2. Patients with histopathologically confirmed diagnosis of renal cell carcinoma
3. Patients with renal cell carcinoma who failed at least one VEGFR TKI
4. Patients with adequate bone marrow function defined as ANC ≥ 1.5 x 109/L, Platelets ≥ 80 x 109/L, Hb >9 g/dL
5. Patients with adequate liver function defined as serum bilirubin ≤ 1.5 x ULN, ALT and AST ≤ 2.5x ULN. Patients with known liver metastases who have an AST and ALT ≤ 5x ULN
6. Patients with adequate renal function defined as serum creatinine ≤ 1.5 x ULN
7. Patients who give a written informed consent obtained according to local guidelines

Exclusion Criteria:

1. CNS disease OR patients with presence or history of central nervous system (CNS) lymphoma
2. Patients receiving chronic, systemic treatment with corticosteroids or another immunosuppressive agent (except corticosteroids with a daily dosage equivalent to prednisone ≤ 20 mg for adrenal insufficiency). However, patients receiving corticosteroids must be on a stable dose for ≥ 4 weeks prior to the first dose of everolimus. Topical or inhaled corticosteroids are permitted.
3. Patients with a known hypersensitivity to everolimus or other rapamycins (sirolimus, temsirolimus) or to its excipients
4. Patients with uncontrolled hyperlipidemia (≥ Grade 3 hyperlipidemia despite optimal supportive medical therapy)
5. Patients with an active, bleeding diathesis
6. Previous organ transplantation
7. Patients who have any severe and/or uncontrolled medical conditions or other conditions that could affect their participation in the study such as:

   * unstable angina pectoris, symptomatic congestive heart failure, myocardial infarction within 6 months of start of study drug, serious uncontrolled cardiac arrhythmia or any other clinically significant cardiac disease
   * severely impaired lung function (spirometry and DLCO that is 50% of the normal predicted value and/or Oxygen saturation that is 88% or less at rest, in room air)
   * uncontrolled diabetes as defined by fasting serum glucose >1.5 x ULN
   * any active (acute or chronic) or uncontrolled infections/disorders
   * non malignant medical illnesses that are uncontrolled or whose control may be jeopardized by the treatment with this study therapy
   * liver disease such as cirrhosis or severe hepatic impairment (Child-Pugh class C).
   * Note: a detailed assessment of Hepatitis B/C medical history and risk factors must be done at screening for all patients. HBV DNA and HCV RNA PCR testing are required at screening for all patients with a positive medical history based on risk factors and/or confirmation of prior HBV/HCV infection.
8. A known history of HIV seropositivity
9. Female patients who are pregnant or breast feeding, or adults of reproductive potential who are not willing to use effective birth control methods. If barrier contraceptives are used, they must be continued throughout the treatment by both sexes.
10. Patients unwilling to or unable to comply with the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2015-09-22 (Actual); Primary Completion 2017-05-05 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
safety and tolerability evaluation (incidence of grade ≥ 2 stomatitis and non-infectious pneumonitis) | up to 36 months
  to evaluate the incidence of grade ≥ 2 stomatitis and non-infectious pneumonitis in RCC patients treated with prednisone 5 mg bid and everolimus 10 mg/day.

SECONDARY OUTCOMES:
Overall response rate (ORR) | up to 36 months
  the sum of partial responses plus complete responses
Progression free survival (PFS) | up to 36 months
  time from the date of starting of the treatment to the date of the first observation of documented disease progression or death due to any cause. Patients without tumor progression at the time of analysis will be censored at their last date of tumor evaluation.
Overall survival (OS) | up to 36 months
  time from the date of starting of the treatment to the date of the death due to any cause. Patients living at the time of analysis will be censored at their last date of tumor evaluation.

CONTACTS AND LOCATIONS:
Overall Officials: Ugo De Giorgi, MD, Principal Investigator — IRST IRCCS, Meldola
Locations (4):
- Italy (4):
  - U.O Oncologia Medica, IRST IRCCS, Meldola, FC
  - Oncologia Medica, PO Faenza, AUSL della Romagna, Faenza, RA
  - Oncologia Medica, PO RAVENNA, AUSL della Romagna, Ravenna, RA
  - Oncologia Medica, PO Rimini-Cattolica, AUSL della Romagna, Rimini

REFERENCES:
- [Derived] Lolli C, Galla V, Schepisi G, Barone D, Burgio SL, Maugeri A, Vertogen B, Amadori D, De Giorgi U. A Phase II Study of Everolimus Plus Oral Prednisone in Patients with Metastatic Renal Cell Cancer. Oncologist. 2017 Jul;22(7):784-e74. doi: 10.1634/theoncologist.2017-0154. Epub 2017 May 25. PMID 28546463